CLINICAL TRIAL: NCT04957238
Title: Impact of a Decision-making Tool to Guide the Use of Physical Restraints in Intensive Care Unit Patients. A Multicentre Randomized Stepped-wedge Trial.
Brief Title: Physical Restraints in Intensive Care Unit Patients
Acronym: ARBORéa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PHRIP 2019 VIDAL
Record Dates: First submitted 2021-03-11; First posted 2021-07-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-09

CONDITIONS: Critically Ill; Intensive Care Unit Delirium; Delirium Confusional State; Agitation,Psychomotor
Keywords: ICU; Physical restraints; Safety; Agitation; Delirium; Nursing care; Sedation; Family; Invasive devices
MeSH Terms: conditions — Critical Illness; Confusion; Psychomotor Agitation; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARBORea decision-making tool (Experimental): After a period of presentation and training on the dedicated decision-making tool (face-to-face, video and paper supports), nurses will be asked to use ARBORéa decision tree. This will be in the form of an electronic file and will give a suggestion of whether or not to use physical restraints. This is based on an algorithm based on specific and mandatory elements (neurological state : RASS (Richmond assessment sedation scale) and CAM-ICU (confusion assessment method-ICU) scores, modification of sedation dosage, equipment levels, presence and adhesion of the family) that will be completed online. ARBORea's suggestion will be collected as well as final caregiver's decision in order to evaluate relevance of the tool. Observations will also be made at least every 8 hours. This period will also be of random duration (stepped wedge)
  Interventions: Other: ARBORea decision-making tool
- Subjective physical restraints use (No Intervention): After study presentation and required data collection description, nurses will complete elements related to ARBORea's tool variables, and inform their actual practices of physical restraints use, at least every 8 hours. ARBORea data concern patient's neurological state (RASS and CAM-ICU scores) and changes in sedation doses. The conditioning will then be filled in to stratify the risk incurred. Pain management will be notified. Finally, the presence and involvement of the families will be collected. Other data, relating to working conditions of the nurses will be collected: nurse to patient ratio, special and time consuming events (new patient admission, in ICU emergencies, need to conduct a patient to CT-scan facility or operative room, change of patient's equipment). Nurse seniority in ICU will be specified. Incidents that have occurred (fall, self-injury, removal of a level C2 equipment). The random duration of this control period will be determined by stepped wedge sequencing.

INTERVENTIONS:
Other: ARBORea decision-making tool — Online ARBORea decision-making tool will guide the use of physical restraints in ICU patients based on objective information on neurological status, level of equipment related to critical illness, and patient's family presence and involvement in patient's surveillance.
  Arms: ARBORea decision-making tool

SUMMARY:
The use of physical restraints is common practice in Intensive Care Units (ICU). This medically prescribed procedure requires full attention of medical and paramedical teams for its implementation, monitoring and ending, as a major restriction of patients' individual freedom. French highest authority for health has defined, for geriatrics and psychiatric units, ten criteria of good practice for physical restraints' use. Routine practice reports critically ill patients' safety as main reason of use. This decision, often left to the sole discretion of nurses, varies according to their own representation of this risk, and depends on several factors: seniority in ICU, nurse to patient ratio and personal workload.

In order to reduce practices subjectivity and heterogeneity, we have developed a decision-making tool for physical restraints implementation. This tool is based on objective scales used on a daily basis concerning neurological status (Richmond Agitation-Sedation Scale (RASS) and Confusion Assessment Method for the ICU (CAM-ICU)). Disorientation or delirium can lead to severe incidents by promoting accidental removing of important devices such as arterial of venous line, drains among others. However, physical restraints are recognized as a major cause of delirium and agitation.

Critically ill patients require rigorous evaluation of organ dysfunctions necessitating adequate invasive equipments, with associated risks of unexpected removal or alteration. Such events could urge caregivers to use physical restraints. Based on recent literature, about a third of ICU patients are restrained, and accidental deconditioning is mainly observed within these particular patients.

In addition, three categories of patients have been defined according to the invasive nature of their equipment and therefore according to the risk associated with an unexpected withdrawal. Finally, presence of patient's family and their adherence to its surveillance were also implemented into the tool. Main study objective is to jointly investigate effectiveness and tolerance of a decision-making tool guiding physical restraints use in ICU patients.

DETAILED DESCRIPTION:
Current study has been designed to measure the impact of an original tool intended to guide the decision to use physical restraints in ICU patients. In a multidisciplinary fashion, we have created a decision-making tool based on objective criteria in an attempt to reduce subjectivity that currently exists in this process of physical restraints use. This tool corresponds to a decision tree based on several criteria:

* the RASS (Richmond Agitation-Sedation Scale) score that assesses patient's state of sedation and agitation. This neurological state could help to determine level of arousal possibly favorizing self-inflicted risks;
* the existence of a delirious state (or delirium), assessed by the CAM-ICU (Confusion Assessment Method for the Intensive Care Unit). This tool is used to detect and assess the presence of a delirium. In the case of a positive CAM-ICU, the patient presents a delirium and may therefore have unsuitable gestures;
* the recent modification of pharmacological-induced sedation allows us to take into account a change in the dosage of infused sedation molecules in order to assess whether the patient may soon find himself in an awakening phase. This transitional phase makes patient's neurological state unstable and can lead to agitation and/or confusion;
* the level of invasive equipment conditioning, defined by the type of device that equips the patient. Three levels of conditioning (C1, C2 and C3) have been defined, ranging from the least to the most harmful in the case of an unexpected removal:

  * Level C1 includes peripheral venous catheters, naso-gastric tubes and urinary catheters;
  * Level C2 includes endotracheal tube, central and arterial lines, renal replacement catheters, drains: thoracic, encephalic or abdominal; intracranial pressure sensors, Swan-Ganz catheters, redons, PICC (peripherally inserted central catheter) lines and Midlines;
  * Level C3 includes veno-venous and veno-arterial ECMO (extra-corporeal membrane oxygenation), intra-aortic counter-pulsion balloons and electro-systolic training probes;
* the presence of patient's family and their adherence to his or her supervision. Families play a key role in patient's care. Their presence might sometimes soothe and reassure the patient. Their adherence and participation to patient's supervision may allow health care team to consider adequate compliance. Regular re-evaluation should then be carried out when they leave patient's room; In order to facilitate the work of caregivers, this decision-making tool has been transcribed into an electronic version that can be accessed online, on a tablet or a computer. Once the above criteria have been filled in, a proposal for whether or not to use physical restraints, as well as main variable criterion for reassessment of this use. This last criterion makes it possible to know the decisive factor that suggested the decision to use restraints or not.

In order to evaluate the impact of this tool on caregivers' decision to use physical restraints, three periods have been planned: a control period in order to evaluate actual practices, a period of training and implementation of the tool, so that each professional is rendered familiar with its use, and finally an intervention period during which the ARBORea tool will be used to suggest physical restraints use.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age, hospitalized in ICU for at least 48 hours.
* Consent to participate in the patient's study or authorization to carry out the research collected from the designated trustworthy person (failing this, a family member, or failing this, a close and stable relation with the person concerned) according to the modalities described in Title II of the book of the First Public Health Code. If no relative is present, the patient may be included on the advice of the investigator (article L. 1111-6). A consent form for continuation of the study and use of the data will then be signed by the patient if and when the patient is again conscious and lucid, or if the patient is unable to express consent, authorization to continue the research will be obtained from the designated trusted person.
* Patient covered by a social security system.

Exclusion Criteria:

* Predictable and uninterrupted maintenance of deep sedation throughout the duration of the stay, due to the seriousness of the lesions, from the moment the patient is admitted to the intensive care unit.
* Lack of predictable remission of a severe coma present on admission to intensive care.
* Refusal to participate by the patient, or by the trusted person contacted by default.
* Patient with DNR (do not resuscitate) orders.
* Patient under legal protection.
* Patient already included in the protocol during another stay in resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Rate of physical restraints use (effectiveness) | Day 0 up to the end of ICU stay, an average of 15 days
  Effectiveness is defined as the rate of observations with the use of restraints; statistical unit will be observations per patient (measured at least every 8 hours) over the entire duration of the ICU stay.
Rate of incidents (tolerance) | Day 0 up to the end of ICU stay, an average of 15 days
  Tolerance is defined as the rate of incidents attributable to non-compliance, corresponding to the deterioration or self-ablation of C2 conditioning, a fall, or self- or hetero-aggressive behaviour. Incidents are determined as soon as an incident occurs, measured every day during ICU stay.

SECONDARY OUTCOMES:
Rate of incidents attributable to physical restraints use | Day 0 up to the end of ICU stay, an average of 15 days
  Deterioration or removal of C2 conditioning, falls, self- or hetero-aggression. As soon as an incident occurs, measured every day during ICU stay.
Rate of incidents without physical restraints use | Day 0 up to the end of ICU stay, an average of 15 days
  Non-restraint incident rates for all levels of conditioning. As soon as an incident occurs, measured every day during ICU stay.
Characteristics of physical restraints | Day 0 up to the end of ICU stay, an average of 15 days
  Typology (upper limbs, lower limbs or abdominal) of the physical restraints performed, in controlled and innovative situations. At least once every 8 hours, during ICU stay, an average of 15 days.
Indications of physical restraints | Day 0 up to the end of ICU stay, an average of 15 days
  Described indications of the physical restraints performed, in controlled and innovative situations. At least once every 8 hours, during ICU stay, an average of 15 days.
Rate of medically prescribed physical restraints | Day 0 up to the end of ICU stay, an average of 15 days
  Number of restraints prescribed in relation to the number of total restraints. At least once every 8 hours, during ICU stay, an average of 15 days.
Characteristics of recorded incidents | Day 0 up to the end of ICU stay, an average of 15 days
  Description of incidents recorded, in controlled and innovative situations. The main types of incidents that can occur are deconditioning, falls, self or hetero aggression. As soon as an incident occurs, measured every day during ICU stay, an average of 15 days.
Rate of recorded incidents | Day 0 up to the end of ICU stay, an average of 15 days
  Rate of incidents recorded, in controlled and innovative situations. The main types of incidents that can occur are deconditioning, falls, self- or hetero-aggressivity, among others. As soon as an incident occurs, measured every day during ICU stay, an average of 15 days.
Short Form Health Survey-36 (SF-36) | Three months after ICU discharge
  Medical outcomes study (SF-36) is a survey that include 36 questions to evaluate patients' quality of life. The result of the questionnaire varies from 0 to 100. A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain.
Impact of Event Scale - Revised (IES-R) | Three months after ICU discharge
  Impact of Event Scale - Revised, is a survey to assess the presence of post-traumatic stress symptoms. It includes 22 items. The total IES-R score is calculated by adding the values obtained for the 22 items (scores 0-88). A score above 22 indicates the presence of acute stress, if the score is above 36 it indicates the presence of post traumatic stress.

CONTACTS AND LOCATIONS:
Overall Officials: Périne Vidal, Principal Investigator — CHU de Clermont-Ferrand
Locations (20):
- France (20):
  - CH Henri Mondor, Aurillac
  - Centre Hospitalier d'Avignon, Avignon
  - Hôpital Nord Franche-Comté, Belfort
  - Centre de Lutte Contre le Cancer Jean-Perrin, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier du Puy en Velay, Le Puy-en-Velay
  - Centre Hospitalier Universitaire - Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon
  - Assistance Publique-Hôpitaux de Marseille - La Timone, Marseille
  - Centre Hospitalier de Montluçon, Montluçon
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Moulins-Yzeure, Moulins
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital de la Pitié Salpétrière, Paris
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier de Salon-de-Provence, Salon-de-Provence
  - CH de Saint Malo, St-Malo
  - Centre Hospitalier Universitaire de Strasbourg - Réa Chirurgicale, Strasbourg
  - Centre Hospitalier Universitaire de Strasbourg -MIR, Strasbourg
  - Centre Hospitalier de Vichy, Vichy

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request, and after steering committee deliberation.

REFERENCES:
- [Derived] Vidal P, Lambert C, Pereira B, Martinez R, Araujo L, Yakhni M, Rolhion C, Morand D, Cosserant S, Genes I, Godet T, Barage A; ARBORea Collaborative group. Stepped wedge cluster randomised controlled trial to assess the impact of a decision support tool for physical restraint use in intensive care units (ARBORea Study): a study protocol. BMJ Open. 2025 May 21;15(5):e085674. doi: 10.1136/bmjopen-2024-085674. PMID 40398949